CLINICAL TRIAL: NCT05063266
Title: Effects of Inspiratory Muscle Training in Pulmonary Hypertensive Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0330 Shaherbano
Record Dates: First submitted 2021-09-13; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Inspiratory Muscle Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Deep Breathing exercise
  Interventions: Other: Deep Breathing Exercise
- Group B (Experimental): Inspiratory Muscle Training
  Interventions: Other: Inspiratory muscle Training

INTERVENTIONS:
Other: Deep Breathing Exercise — control groups received deep breathing exercise 6 days a week for two weeks. Deep breathing exercises includes diaphragmatic breathing and pursed lip breathing.
  Arms: Group A
Other: Inspiratory muscle Training — Treatment group received inspiratory muscle training 20 minutes 6 days a week for two weeks.IMT was done by using pressure threshold device.
  Arms: Group B

SUMMARY:
Although the progressive nature of pulmonary hypertension (PH), including the impairment of respiratory muscle function, studies have demonstrated beneficial effects of physical exercise on the functional limitations caused by the disease in this population, being an important collaborator to the conventional drug therapy.Respiratory muscle training (RMT) improves functional capacity and quality of life (QoL) in patients.A randomized controlled trial was conducted to evaluate the effectiveness of this protocol on respiratory muscle strength and endurance, functional capacity. 18 subjects were allocated in 2 groups, group A was control group and group B was experimental group. Group A or Control group received deep breathing exercises. Group B received 30 minutes of IMT 6days weekly for 2 weeks by using a pressure threshold device. The purpose of this study was to investigate the effects of inspiratory muscle training (IMT) in PAH. To evaluate effectiveness of IMT mouth pressure device ,functional capacity using 6 minute walking test (6MWT)health assessment via SF 36 questionnaire were used before and after training protocol.

ELIGIBILITY:
Inclusion Criteria:

Age group of 40 to 70 years.

* Both male and females will be included.
* Patients with a diagnosis of PH (PAPm ≥ 25mmHg and PAOP <15mmHg);
* Clinically stable with augmented and unchanged daily medication therapy in the last three months; Subjects who agree to contribute in the research by signing a free and knowledgeable consent form.

Exclusion Criteria:

* COPD
* Severe ischemic heart disease
* Left heart failure;
* Cor pulmonale
* Cognitive disorders;
* Orthopedic problems; e.g;fracture in thoracic region.
* Emergency or elective surgical intervention during the protocol;
* Recent viral infections;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
6-min walk test (6 MWT) | 2nd week
  The 6-min walk test (6 MWT) is a submaximal exercise test drive that includes measurement of distance walked throughout a period of 6 minutes. The 6-minute walk distance (6 MWD) stipulates a measure for collective global retort of multiple cardiopulmonary and musculoskeletal structures involved in workout.The 6 MWT provides information about functional capacity, response to rehabilitation and prognosis slanting a broad range of chronic cardiopulmonary situations. Main strengths of the 6 MWT curb from its simplicity in conception and performing, low cost, ease of consistency, and acceptance by test individuals, including those who are deconditioned, aged, or fragile.
SF 36 | 2nd week
  SF-36 is a setting of universal, clear, and easily instructed quality-of-life methods. These measures hang on upon patient self-reporting and are now widely utilized by trained care groups and by Medicare for everyday observing and assessment of care findings in mature patient role

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha kausar, PP-DPT, Study Chair — Riphah International University
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan P, Yuan XT, Sun XY, Pudasaini B, Liu JM, Hu QH. Exercise training for pulmonary hypertension: a systematic review and meta-analysis. Int J Cardiol. 2015 Jan 15;178:142-6. doi: 10.1016/j.ijcard.2014.10.161. Epub 2014 Oct 27. No abstract available. PMID 25464238
- [Background] Chia KS, Wong PK, Faux SG, McLachlan CS, Kotlyar E. The benefit of exercise training in pulmonary hypertension: a clinical review. Intern Med J. 2017 Apr;47(4):361-369. doi: 10.1111/imj.13159. PMID 27338855
- [Background] Becker-Grunig T, Klose H, Ehlken N, Lichtblau M, Nagel C, Fischer C, Gorenflo M, Tiede H, Schranz D, Hager A, Kaemmerer H, Miera O, Ulrich S, Speich R, Uiker S, Grunig E. Efficacy of exercise training in pulmonary arterial hypertension associated with congenital heart disease. Int J Cardiol. 2013 Sep 20;168(1):375-81. doi: 10.1016/j.ijcard.2012.09.036. Epub 2012 Oct 5. PMID 23041100
- [Background] Saglam M, Arikan H, Vardar-Yagli N, Calik-Kutukcu E, Inal-Ince D, Savci S, Akdogan A, Yokusoglu M, Kaya EB, Tokgozoglu L. Inspiratory muscle training in pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2015 May-Jun;35(3):198-206. doi: 10.1097/HCR.0000000000000117. PMID 25909652
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284